CLINICAL TRIAL: NCT03158506
Title: An Open-Label, Single Center Study to Assess the Absorption, Metabolism, Excretion, and Mass Balance of a Single Oral Dose of 50 mg (90 uCi) [14C]-HMS5552 in Healthy Adult Male Subjects
Brief Title: Human Mass Balance Study of HMS5552 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMM0105
Record Dates: First submitted 2017-05-10; First posted 2017-05-18 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2017-04

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Dorzagliatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [C14]-labelled HMS5552 (Experimental)
  Interventions: Drug: HMS5552

INTERVENTIONS:
Drug: HMS5552 — [14C]-labelled HMS5552

SUMMARY:
This is an open-label, single center, 1-period study in healthy adult male subjects to assess absorption, metabolism, and excretion of HMS5552 after a single oral administration of 50 mg (90 μCi) of [14C]-HMS5552.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male 19-55 years of age
* Weight at least 50 kg, and BMI within the range of 18-30 kg/m2
* Written informed consent must be obtained before any assessment is performed

Exclusion Criteria:

* History or presence of clinically significant medical, surgical or psychiatric condition or disease in the opinion of the Investigator or designee which might significantly alter the absorption, distribution, metabolism and excretion of drugs.
* History or presence of alcoholism or drug abuse.
* Smoker.
* Abnormal bowel habits.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
Total radioactivity in blood, plasma urine and feces | Up to 168 hours
  Peak plasma concentration (Cmax)
Total radioactivity in blood, plasma urine and feces | Up to 168 hours
  Area under the plasma concentration versus time curve (AUC)
Total radioactivity in blood, plasma urine and feces | Up to 168 hours
  Time to reach Cmax (Tmax)
Total radioactivity in blood, plasma urine and feces | Up to 168 hours
  Total radioactivity in urine and faeces at each time interval and cumulative radioactivity (mass balance)

SECONDARY OUTCOMES:
Concentrations of HMS5552 and its metabolites in plasma, urine and feces | Up to 168 hours
  Peak plasma concentration (Cmax)
Number of participants with adverse events as a measure of safety and tolerability | Up to 168 hours
  Adverse events; Laboratory parameters; Vital signs, clinical signs and symptoms and physical examination, including changes from baseline; ECG evaluation
Concentrations of HMS5552 and its metabolites in plasma, urine and feces | Up to 168 hours
  Area under the plasma concentration versus time curve (AUC)
Concentrations of HMS5552 and its metabolites in plasma, urine and feces | Up to 168 hours
  Time to reach Cmax (Tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Tomek, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No